CLINICAL TRIAL: NCT01756378
Title: Effect of Mulligan'Mobilization With Movement on Pain, Disability and Range of Motion in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Magdolin Mishel Samy Saad Shenouda, lecturer of physical tehrapy for musc uloskeletal disorders, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/012/003
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Physical Fittness
Keywords: Mobilization with movement,knee osteoarthritis,
MeSH Terms: interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Muligan mobilization with movement (Experimental): Interventions are:
  medial glide mobilization with movement lateral glide mobilization with movement rotation mobilization with movement dorsal glide with active knee flexion
  Interventions: Procedure: joint mobilization with movement; Procedure: traditional physical therapy program
- traditional physical therapy program (Active Comparator): Infra-red, stretching exercises, strengthening exercises,
  Interventions: Procedure: traditional physical therapy program

INTERVENTIONS:
Procedure: joint mobilization with movement
  Other Names: Muligan's technique
  Arms: Muligan mobilization with movement
Procedure: traditional physical therapy program — I.R, stretching exercises, strengthen exercises

SUMMARY:
we tested the effect of adding the mobilization with movement to the traditional physical therapy program on pain, ROM and functional disability in patients with knee OA.

study hypothesis: there will be no significant difference between traditional physical therapy program and the mobilization with movement plus the traditional physical therapy program on pain, ROM and functional disability in patients with knee OA

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral osteoarthritis knee age ranges from 30-60 years old grade 1 or 2 on Kallegren and Lawerance scale. body mass index not more than 36

Exclusion Criteria:

* history of major knee injury or surgery, tumors, osteoporosis, patients undertaking analgesics, patients with uncontrolled hypertension, bleeding, dermatological problems, psychiatric disorders, hearing problems, cognitive problems and pacemaker.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
pain | baseline and up to 10 months
  measured by visual analogue scale
functional disability | baseline and up to 10 months
  measured by WOMAC scale
Range of motion for the knee joint | baseline and up to 10 months
  measured by Gynom digital electrogoniometer

CONTACTS AND LOCATIONS:
Overall Officials: Magdolin M Shenouda, Ph.D, Study Director — Faculty of Physical Therapy, Cairo Un iversity; Reda K Gad ElHak, Ms.C, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt